CLINICAL TRIAL: NCT00617942
Title: BrUOG-BR-211B q3week Carboplatin With Weekly Abraxane and Trastuzumab As Neoadjuvant Therapy in Resectable and Unresectable HER2+ (Stage IIa-IIIb) Breast Cancer
Brief Title: Neoadjuvant Carboplatin, Weekly Abraxane and Trastuzumab in HER2+ Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: William Sikov MD (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor-Investigator, William Sikov MD, Principle Investigator, Brown University
Organization: Brown University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-BR-211B
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Results first posted 2017-08-22 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Trastuzumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Neo-adjuvant cohort 1 (Experimental)
  Interventions: Drug: Cohort 1 neo-adjuvant
- Neo-adjuvant cohort 2 (Experimental)
  Interventions: Drug: Cohort 2 neo-adjuvant
- Adjuvant cohort 1 (Experimental)
  Interventions: Drug: Cohort 1 adjuvant
- Adjuvant cohort 2 (Experimental)
  Interventions: Drug: Cohort 2 adjuvant

INTERVENTIONS:
Drug: Cohort 1 neo-adjuvant — Cohort 1 : Trastuzumab 6 mg/kg IV over 60 minutes day -14
  Trastuzumab 2 mg/kg IV over 60 minutes weekly then Abraxane 100 mg/m2 IV over 30 minutes weekly x 18 weeks followed by Carboplatin at AUC 6 IV over 30 min weeks 1,4,7,10,13 and 16
  Other Names: Abraxane (nab-paclitaxel), Herceptin (trastuzumab) and carboplatin
  Arms: Neo-adjuvant cohort 1
Drug: Cohort 2 neo-adjuvant — Cohort 2 :Abraxane 100 mg/m2 IV over 30 minutes days -14 and -7 Trastuzumab 2 mg/kg IV over 60 minutes weekly (4 mg/kg week 1) then Abraxane 100 mg/m2 IV over 30 minutes weekly x 18 weeks followed by Carboplatin at AUC 6 IV over 30 min weeks 1,4,7,10,13 and 16
  Arms: Neo-adjuvant cohort 2
Drug: Cohort 1 adjuvant — Trastuzumab 8 mg/kg x 1 dose, then 6 mg/kg q3wks x 11 doses Adjuvant chemotherapy, post-op radiation and hormonal therapy at discretion of treating physicians
  Arms: Adjuvant cohort 1
Drug: Cohort 2 adjuvant — Trastuzumab 8 mg/kg x 1 dose, then 6 mg/kg q3wks x 11 doses Adjuvant chemotherapy, post-op radiation and hormonal therapy at discretion of treating physicians
  Arms: Adjuvant cohort 2

SUMMARY:
Q3week carboplatin with weekly abraxane and trastuzumab as neoadjuvant therapy in resectable and unresectable HER2+ (stage IIa-IIIb) breast cancer

DETAILED DESCRIPTION:
Our goal is to develop an induction chemotherapy regimen that will have a pCR rate above 50% in HER2+ patients without exposing patients to the toxicity of an anthracycline-based regimen. A minimum of 60 evaluable patients will be accrued to the study. We are assuming an observed pCR (or near pCR) rate of 70%. Assuming no more than 10% of patients will be inevaluable for the primary endpoint (pCR), we will have at least 54 evaluable patients. With this number, we will have 90% power, with a 1-sided alpha error of 0.05, to demonstrate a pCR rate exceeding 50% for our novel regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the breast
* ANC > 1000 cells
* Female; age > 18; Zubrod PS 0-1
* Platelets > 100,000
* Stage IIA-IIIB disease
* Total bilirubin < or = ULN
* No evidence of metastatic disease Not pregnant or lactating
* No prior systemic therapy for this breast cancer
* Serum Creatinine < 1.5 mg/dl or Creat Cl > 30 ml/min
* Serum ALT < 2.5 x ULN
* ER, PR and HER2 status required
* LVEF (MUGA/echo)WNL
* No baseline > 2 neuropathy
* Hemoglobin > 9.0 gm/dl
* HER2+, defined by IHC 3+ or FISH ratio > 2.0

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2012-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Sikov, MD, Principal Investigator — Brown University
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Yale Smilow Cancer Center, New Haven, Connecticut
  - Women and Infants Hospital, Providence, Rhode Island
  - Roger Williams Medical Center, Providence, Rhode Island
  - Rhode Island and The Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Cheng H, Bai Y, Sikov W, Sinclair N, Bossuyt V, Abu-Khalaf MM, Harris LN, Rimm DL. Quantitative measurements of HER2 and phospho-HER2 expression: correlation with pathologic response to neoadjuvant chemotherapy and trastuzumab. BMC Cancer. 2014 May 8;14:326. doi: 10.1186/1471-2407-14-326. PMID 24885187

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Cohort 1 neo-adjuvant: Cohort 1 : Trastuzumab 6 mg/kg IV over 60 minutes day -14
  Trastuzumab 2 mg/kg IV over 60 minutes weekly then Abraxane 100 mg/m2 IV over 30 minutes weekly x 18 weeks followed by Carboplatin at AUC 6 IV over 30 min weeks 1,4,7,10,13 and 16
  Cohort 1 adjuvant: Trastuzumab 8 mg/kg x 1 dose, then 6 mg/kg q3wks x 11 doses Adjuvant chemotherapy, post-op radiation and hormonal therapy at discretion of treating physicians
- Cohort 2: Cohort 2 neo-adjuvant: Cohort 2 :Abraxane 100 mg/m2 IV over 30 minutes days -14 and -7 Trastuzumab 2 mg/kg IV over 60 minutes weekly (4 mg/kg week 1) then Abraxane 100 mg/m2 IV over 30 minutes weekly x 18 weeks followed by Carboplatin at AUC 6 IV over 30 min weeks 1,4,7,10,13 and 16
  Cohort 2 adjuvant: Trastuzumab 8 mg/kg x 1 dose, then 6 mg/kg q3wks x 11 doses Adjuvant chemotherapy, post-op radiation and hormonal therapy at discretion of treating physicians
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 37 | 23
Completed | 29 | 19
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 37 | 23 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 20 | 54
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 51.4 [32 to 72] | 51.6 [35 to 70] | 51.5 [32 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 23 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 23 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Pathologic Response Rate, Observed Following Treatment With q3week Carboplatin, Weekly Abraxane and Weekly Trastuzumab in Resectable and Unresectable LABC;
Description: These numbers represent patients with a RCB score of zero (0). RCB stands for residual cancer burden.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 37 | 23
participants | 12 | 13

2. Secondary Outcome: Patients Affected by Toxicities of Regimen During Treatment, Including Grade >2 Neurotoxicity the Incidence of Subclinical and Clinical Cardiac Toxicity
Description: Please note that these events represent toxicities that were experienced during treatment, but that does not mean that all toxicities were indeed deemed related to study treatment.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Neo-adjuvant Cohort 1 | Neo-adjuvant Cohort 2 | Adjuvant Cohort 1 | Adjuvant Cohort 2
Number analyzed (Participants) | 37 | 23 | 29 | 19
participants | 37 | 23 | 29 | 19

ADVERSE EVENTS:
Time Frame: Toxicities were captured at start of treatment through 1 year of adjuvant trastuzumab. CTCAE version 3.0 was used.
Description: Please note that all AEs are reported here but this does not mean that all toxicities were deemed related to study treatment.
Arm/Group | Neo-adjuvant Cohort 1 | Neo-adjuvant Cohort 2 | Adjuvant Cohort 1 | Adjuvant Cohort 2
Serious Adverse Events (participants affected / at risk) | 7/37 | 8/23 | 5/29 | 3/19
Other Adverse Events (participants affected / at risk) | 37/37 | 23/23 | 29/29 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neo-adjuvant Cohort 1 (N=37) | Neo-adjuvant Cohort 2 (N=23) | Adjuvant Cohort 1 (N=29) | Adjuvant Cohort 2 (N=19)
gr 3port infection, (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
flu (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile Neutropenia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gr 4 sepsis, intubated (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — neutro 3, anemia 3, thromb 4, HTN 4, arf 3, hypok 4, hypocal 4, ards 4, hyperbili 3, tach 4, fever 2
Diarrhea gr 2, Nausea gr 3, infection gr 3 (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
infection normal ANC/viral grade 1 (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration 3, Diarrhea 3, Vomit 3, HGB3, Nausea 3, K 3, Dyspnea 2 (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gr 3cellulitis - breast (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
gr 3 diarrhea, gr 2 neutropenia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UTI, gr 3 ANC, gr 3 HGB, Gr3 infection, Gr 2 fever and pain, gr1 rigor (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
fever unknown etiology gr 1, lymphatics gr 1 (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncopal epidose gr 3, dehydration gr 2, diabetes gr 2, anemia gr 2 (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
thrombus occlusive L IJ gr 3, hypomagnesia gr 1, hypokalemia gr 1 (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dehydr gr3, chest pain gr 3, (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hypotension gr 2, HGB gr 3, Fever gr2, creatinine gr 1, diarrhea gr 2, infection gr 3, ANC gr 3,
gr 3 left jugular thrombis , anemia gr 2, (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
left ear otitis externa gr 3, ANC 4, WBC 2 Diarrhea 1 (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
vomit gr 3, Nausea gr 3, diarrhea gr2, GI bleed gr 2, Abdominal pain rg3, (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — hgb gr 2, Na 1, K 1, Ca 1, ANC 2, Anorexia 3,dehydration gr3, cr gr 1, WBC gr 2,
vomiting gr 3, infection Cdiff gr 3, Hypokalemia gr 1, gr 1 hypomagnesia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
right upper extremity cellulitis gr 3, (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — right ue pain gr 2, UTI gr 2, WBC gr 2, HGB gr 2, ANC gr 2, K gr 2, hypoalbum gr 1, INR gr 1, constipation gr 1,
gr 3 ulcerative colitis exacerbation with and without gr 1 fever) (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
gran mal seizure-2 (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
allergic rxn (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia gr 2, Anemia 2, ANC 4, (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — External ear inflammation 1, tachycardia 1, PLT 1, Myalgias 2
suicidal ideation gr 2 and depression gr 3 not related (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
post re-construction pt experienced seroma grade 2 (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hernia grade 3 secondary to surgery healing issue (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis 3, PLT 1, K, 1, Ca, 1, Hgb1, Phos, 3, Pruritis, 1 (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cardiac ischemia gr 2, (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
gr 3 abd pain, gr 1 nausea, gr 2 vomitting (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
impt medical event(gr2) abnormal stress test need for cardiac cath (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neo-adjuvant Cohort 1 (N=37) | Neo-adjuvant Cohort 2 (N=23) | Adjuvant Cohort 1 (N=29) | Adjuvant Cohort 2 (N=19)
WBC (Investigations) | 32 (32) | 21 (21) | 12 (12) | 9 (9)
ANC (Investigations) | 32 (32) | 19 (20) | 7 (7) | 4 (4)
plt (Investigations) | 33 (33) | 20 (20) | 6 (6) | 4 (4)
HGB (Investigations) | 35 (35) | 22 (22) | 23 (23) | 12 (12)
M/A (Investigations) | 10 (10) | 9 (9) | 4 (4) | 4 (4)
creatinine (Investigations) | 7 (7) | 3 (3) | 0 (0) | 2 (2)
Anorexia (Investigations) | 5 (5) | 11 (11) | 0 (0) | 7 (7)
wt loss (Investigations) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Fatigue (Investigations) | 28 (28) | 21 (21) | 16 (16) | 14 (14)
Rash (Investigations) | 3 (3) | 15 (15) | 6 (6) | 11 (11)
nausea (Investigations) | 21 (21) | 18 (18) | 2 (2) | 10 (10)
vomiting (Investigations) | 6 (6) | 6 (6) | 2 (2) | 3 (3)
mucositis (Investigations) | 6 (6) | 9 (9) | 0 (0) | 5 (5)
diarrhea (Investigations) | 8 (8) | 17 (17) | 4 (4) | 7 (7)
rhinitis (Investigations) | 0 (0) | 13 (13) | 0 (0) | 9 (9)
AST/ALT (Investigations) | 28 (28) | 9 (9) | 11 (11) | 6 (6)
Neurosensory (Investigations) | 11 (11) | 20 (20) | 4 (4) | 17 (17)
Neuromuscular (Investigations) | 9 (9) | 7 (7) | 4 (4) | 9 (9)
(Investigations) | 6 (6) | 2 (2) | 2 (2) | 1 (1)
K (Investigations) | 12 (12) | 8 (8) | 4 (4) | 6 (6)
Mg (Investigations) | 20 (20) | 7 (7) | 6 (6) | 5 (5)
Ca (Investigations) | 7 (7) | 7 (7) | 4 (4) | 7 (7)
Phos (Investigations) | 4 (4) | 4 (4) | 4 (4) | 1 (1)
Infection (Investigations) | 6 (6) | 6 (6) | 1 (1) | 7 (7)
HTN (Investigations) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Abd pain (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
tinnuitius (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
cough (Investigations) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
chest pain (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
epistaxis (Investigations) | 1 (1) | 5 (5) | 0 (0) | 3 (3)
pulmonary embolism (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
wt gain (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
ocular (Investigations) | 0 (0) | 4 (4) | 1 (1) | 4 (4)
rectal bleed (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
insomnia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
glucose (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dyspnea (Investigations) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
alopecia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
heartburn (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
rigors (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
edema (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dizziness (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
headache (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
troponin (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
tachycardia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hyperpigmentation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
proteinuria (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SOB (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
desquam skin (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
back pain (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
glucose (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DVT (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pain breast (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
mood alteration (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
chelitis (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
albumin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hypouricemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No